CLINICAL TRIAL: NCT05642208
Title: Dupilumab Step-down Strategy to Maintain Remission in Adult and Adolescents Patients With Atopic Dermatitis: a Non-inferiority Randomized Trial
Brief Title: Dupilumab Step-down Strategy to Maintain Remission in Adult and Adolescents Patients With Atopic Dermatitis
Acronym: MADULO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0378
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis; Eczema, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Injections will be spaced as :
  * Every 3 weeks between M0 and M4,
  * Every 4 weeks between M4 and M8 (if ADCT<7 and IGA ≤ 2, AD assessed as controlled by the investigator and stable amount of local treatment used),
  * Then every 5 weeks until the end of the clinical trial (M12) (if ADCT<7 and IGA ≤ 2, AD assessed as controlled by the investigator and stable amount of local treatment used).
  In case of ADCT≥7 or IGA > 2 or disease assessed as uncontrolled by the investigator, the injection interval treatment will be step up to the previous interval.
  The treatment is administered subcutaneously and can be delivered in pen or syringe for subcutaneous injection.
  The dosage is usually :
  * 300 mg per injection for adults and adolescents (12-17 years) weighing more than 60 kg
  * 200 mg per injection for adolescents (12-17 years) weighing less than 60 kg.
  Interventions: Drug: Dupilumab step-down
- Control group (No Intervention): in this group the interval between injections is maintained every 2 weeks (14 days) throughout the clinical trial.
  The treatment is administered subcutaneously and can be delivered in pen or syringe for subcutaneous injection.
  Treatment will be prescribed in the control group according to the marketing authorization dosage (see paragraph 5.1). The dosage is usually :
  * 300 mg every 14 days for adults and adolescents (12-17 years) weighing more than 60 kg
  * 200 mg every 14 days for adolescents (12-17 years) weighing less than 60 kg.

INTERVENTIONS:
Drug: Dupilumab step-down — step down dupilumab injections
  Arms: Experimental Group

SUMMARY:
The goal of this clinical trial is to compare a step-down strategy of spacing dupilumab injections with a standard maintenance treatment in adolescents and adults with controlled Atopic dermatitis (AD) for at least six months. The impact of dosage reduction strategies will be assessed with an innovative primary endpoint: the area under the curve of the weekly ADCT assessment.

DETAILED DESCRIPTION:
For both groups:

At inclusion visit :

* Patient information and signature of consent form
* Randomisation
* Previous medical history
* Clinical exam
* Recording ADCT, EASI, IGA, NRS pruritus, DLQI or CDLQI, EQ-5D-5L

Weekly during 12 months (by patients on https://hestia.chu-nantes.fr) :

* Self-assessment of ADCT
* Date of dupilumab injections
* Batch number of dupilumab
* Amount of topical corticosteroids

Visits at M4, M8 and M12 will be performed for :

* Clinical exam
* Recording secondary end points (EASI, IGA, NRS pruritus, DLQI or CDLQI, EQ-5D-5L) and adverse events
* Collect out-of-pocket expenses (M4 and M12).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* Moderate to severe AD treated with dupilumab every 2 weeks
* Written informed consent (patient and/or person who has parental authority)
* Dupilumab treatment for at least one year
* Controlled AD (ADCT<7 and IGA ≤ 2) and assessed as controlled by the investigator since at least 6 months without tapering dosage of dupilumab
* Amount of topical treatment (TCS or calcineurin inhibitor) stable for 6 months and less than 60 g/month

Exclusion Criteria:

* Patients with Side effects of dupilumab
* Non controlled AD: ADCT ≥ 7 or IGA ≥ 3
* Female patient must not be pregnant*, breastfeeding or considering becoming pregnant
* Patient under judicial protection
* Adults under guardianship or trusteeship

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of Atopic Dermatitis Control Tool (ADCT) | over 12 months
  to demonstrate the non-inferiority of a step down dosage strategy of dupilumab as compared with maintenance of initial treatment, on long-term control of the disease severity at one year in adolescents and adults patients with controlled AD.The primary endpoint is the Area under the curve of Atopic Dermatitis Control Tool (ADCT) score achieved by the patient every week during one year.
  As the ADCT score refers to the last 7 days, a weekly assessment is the most accurate to detect all variations in disease severity intensity.

SECONDARY OUTCOMES:
Mean difference in EASI score | every 4 months over 12 months
  to assess the efficacy of a tapering dosage strategy of dupilumab among patients (adolescents from 12 years old and adults) with controlled AD as compared to the standard maintenance strategy on the Eczema Area and Severity Index Mean difference in EASI score from baseline to month 4, month 8, month 12(EASI)
Mean difference in Investigator global assessment | every 4 months over 12 months
  to assess the efficacy of a tapering dosage strategy of dupilumab among patients (adolescents from 12 years old and adults) with controlled AD as compared to the standard maintenance strategy on the Investigator Global assessment (IGA) Mean difference in Investigator global assessment from baseline to month 4, month 8, month 12
Mean difference in Itch numerical rating scale | every 4 months over 12 months
  to assess the efficacy of a tapering dosage strategy of dupilumab among patients (adolescents from 12 years old and adults) with controlled AD as compared to the standard maintenance strategy on the Itch numerical rating scale Mean difference in Itch numerical rating scale from baseline to month 4, month 8, month 12
The patient quality of life will be assessed with the DLQI (Dermatology Life Quality Index) measured at M4, M8, M12 or with the CDLQI (Children Dermatology Life Quality Index) for children under 16. Mean difference in DLQI (CDLQI for children <16) | every 4 months over 12 months
  The patient quality of life will be assessed with the DLQI (Dermatology Life Quality Index) measured at month 4, month 8, month 12 or with the CDLQI (Children Dermatology Life Quality Index) for children under 16. Mean difference in DLQI (CDLQI for children <16) from baseline to month 4, month 8, month 12 will be assessed.
  to assess the efficacy of a tapering dosage strategy of dupilumab among patients (adolescents from 12 years old and adults) with controlled AD as compared to the standard maintenance strategy on the patient quality of life.
cost-utility analysis performed from a health care system perspective | over 12 months
  The economic efficiency will be assessed by a cost-utility analysis performed from a health care system perspective (i.e. considering only direct health care costs) and a 1-year time horizon. Incremental cost-utility ratio (cost per Quality-Adjusted Life-Years, QALYs) from a health care system perspective and with a 1-year time horizon will be taken into account.
  to assess the efficacy of a tapering dosage strategy of dupilumab among patients (adolescents from 12 years old and adults) with controlled AD as compared to the standard maintenance strategy on the economic efficiency
Incremental cost-utility ratio (cost per Quality-Adjusted Life-Years, QALYs) from a health care system perspective | over 12 months
  The economic efficiency will be assessed by a cost-utility analysis performed from a health care system perspective (i.e. considering only direct health care costs) and a 1-year time horizon. Incremental cost-utility ratio (cost per Quality-Adjusted Life-Years, QALYs) from a health care system perspective and with a 1-year time horizon will be taken into account.
  to assess the efficacy of a tapering dosage strategy of dupilumab among patients (adolescents from 12 years old and adults) with controlled AD as compared to the standard maintenance strategy on the economic efficiency

CONTACTS AND LOCATIONS:
Overall Officials: Hélène AUBERT, Principal Investigator — Nantes University Hospital
Locations (32):
- France (31):
  - Amiens University hospital, Amiens
  - CHU d'Angers, Angers
  - Hôpital Victor Dupouy, Argenteuil
  - CHU de Besançon, Besançon
  - CHU de Bordeaux Adulte, Bordeaux
  - CHRU de Brest, Brest
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - GH La Rochelle - Ré-Aunis, La Rochelle
  - CH de Le Mans, Le Mans
  - CHRU de Lille, Lille
  - Groupement des Hôpitaux de l'institut Catholique de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital de la Timone, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CH de Niort, Niort
  - Hôpital Cochin, Paris
  - Hôpital Necker-Enfants malades, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Tenon, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CH de Saint Nazaire, Saint-Nazaire
  - HIA Sainte Anne, Toulon
  - CHU de Toulouse - Hôpital Larrey, Toulouse
  - CHRU de Tours, Tours
- CHU de La Réunion, Saint-Pierre, La Réunion, Reunion

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Foureau A, Faurel-Paul E, Hardouin JB, Papinot L, Schirr-Bonnans S, Tessier P, Jobert A, Poinas A, Staumont-Salle D, Tauber M, Chosidow O, Barbarot S, Aubert H; the FRench Atopic DErmatitis Network from de GREAT Research group. Dupilumab step-down strategy to maintain remission in adult and adolescent patients with atopic dermatitis: study protocol for a non-inferiority randomized trial (MADULO). Trials. 2025 Dec 5;27(1):26. doi: 10.1186/s13063-025-09325-4. PMID 41350756